CLINICAL TRIAL: NCT04166123
Title: Psychometric Properties of the Elderly Health Questionnaire in Frailty Risk Assessment Among Community-dwelling Older People
Brief Title: Psychometric Properties of the Elderly Health Questionnaire Among Community-dwelling Older People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901045RINA
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Frailty
Keywords: frailty; older adults; instrument; community
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study are to validate the reliability and validity of Elderly Health Questionnaire in assessing frailty risk of community-dwelling older adults.

DETAILED DESCRIPTION:
The aims of this study are to validate the test-retest reliability, internal consistency, criterion-related validity, predictive validity and construct validity of Elderly Health Questionnaire in assessing frailty risk of community-dwelling older adults.

The investigators conduct a prospective study to require data of health states, function, lifestyle and quality of life in community-dwelling older adults ,and will recruit about 150 subjects in NTUH and communities in Taipei City. The investigators analyze the (change) scores of Elderly Health Questionnaire to test the internal consistency and test-retest reliability. Also, the investigators test the correlation between the scores of Elderly Health Questionnaire and the scores of the other measurements (i.e., HELP-T, WHOQOL-BREF, MoCA, SPPB, UPSA-B) to validate the concurrent validity, and the correlation between the scores of Elderly Health Questionnaire and the scores of CFS to validate predictive validity. The construct validity is validated by exploratory factor analysis.

ELIGIBILITY:
Inclusion Criteria:

* aged > 65 years old
* able to read
* Clinical frailty scale ≦ 6

Exclusion Criteria:

* diagnosed as dementia or schizophrenia
* active cancer receiving treatment
* terminal cancer patient
* hospitalization in 1 month
* with implantable device
* couldn't follow the instructions
* wheelchair bound

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: over 65 years old community-dwelling elderly
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Elderly Health Questionnaire | an average of 2-4 weeks between pretest and posttest (baseline, week 2-4)
  It is a self-report questionnaire about frailty and health conditions. Each item is scored 0 or 1, yielding a total of 0-70. The scores range from 0 (best performance) to 70 (worst performance).

SECONDARY OUTCOMES:
Taiwanese version of the Health Enhancement Lifestyle Profile (HELP-T) | pretest (baseline)
  HELP-T is a 59-item self-report questionnaire measuring various aspects of health-related lifestyles in older adults. The scores range from 0 (worst performance) to 118 (best performance).
WHOQOL-BREF Taiwan version | pretest (baseline)
  It is a cultural-specific self-report questionnaire measuring health-related quality of life in Taiwan. The scores range from 0 (worst QoL) to 100 (best QoL).
Short physical performance battery (SPPB) | pretest (baseline)
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 4 (best performance).
Montreal Cognitive Assessment (MoCA) | pretest (baseline)
  The MoCA is a cognitive screening test designed to assist health professionals in the detection of mild cognitive impairment and Alzheimer's disease. The MoCA Test was validated in the setting of mild cognitive impairment (MCI), and has been subsequently adopted in numerous clinical settings. The sensivity of the MoCA for detecting MCI is 90%, compared to 18% for other leading cognitive screening tools such as the MMSE. The scores range from 0 (worst performance) to 30 (best performance).
Brief University of California at San Diego Performance-Based Skills Assessment (UPSA-B) | pretest (baseline)
  UPSA-B is a shorter version of the UPSA-2 that uses only the financial skills and communication skills subscales (i.e. counting change, telephone calls, and paying bills). This version of the UPSA takes approximately 15 minutes to complete and has been shown to be an accurate predictor of patient ability to live independently, as compared to the full version of the UPSA. The scores range from 0 (worst performance) to 20 (best performance).
Canadian Study of Health and Aging Clinical Frailty Scale (CFS) | pretest (baseline)
  CFS is a frailty tool derived using data from the Canadian Study of Health and Aging, a national 5-year prospective cohort study. The CFS is a judgment-based scale that considers clinical data on a patient's cognition, mobility, function, and comorbidities. The scores range from 1 (very fit) to 9 (terminally ill).

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, MS, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan